CLINICAL TRIAL: NCT01683409
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging, Phase 2 Study to Evaluate the Safety and Renal Efficacy of Baricitinib in Patients With Diabetic Kidney Disease
Brief Title: A Study to Test Safety and Efficacy of Baricitinib in Participants With Diabetic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14734; I4V-MC-JAGQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Administered orally, given as three placebo tablets in the morning and one placebo tablet in the evening for 24 weeks.
  Interventions: Drug: Placebo
- Baricitinib 0.75 mg/0.5 mg QD (Experimental): Administered orally, 0.75 mg given as one 0.75 mg tablets and two placebo tablets in the morning and one placebo tablet in the evening for 24 weeks or 0.5 mg given as one 0.5 mg tablet and two placebo tablets in the morning and one placebo tablet in the evening for 24 weeks. Placebo tablets given to maintain blind.
  Interventions: Drug: Baricitinib; Drug: Placebo
- Baricitinib 0.75 mg/0.5 mg BID (Experimental): Administered orally, 0.75 mg given as one 0.75 tablet and 2 placebo in the morning and one 0.75 mg tablet in the evening for 24 weeks or 0.5 mg given as one 0.5 mg tablet and two placebo tablets in the morning and one 0.5 mg tablet in the evening. Placebo tablets given to maintain blind.
  Interventions: Drug: Baricitinib; Drug: Placebo
- Baricitinib 1.5 mg/1 mg (Experimental): Administered orally, 1.5 mg given as two 0.75 mg tablets and 1 placebo tablet in the morning and one placebo tablet in the evening for 24 weeks or 1 mg tablet and two placebo tablets in the morning and one placebo tablet in the evening for 24 weeks. Placebo tablets given to maintain blind.
  Interventions: Drug: Baricitinib; Drug: Placebo
- Baricitinib 4 mg/2.75 mg (Experimental): Administered orally, 4 mg given as one tablet and 2 placebo tablets in the morning and one placebo tablet in the evening for 24 weeks or 2.75 mg given as two 1 mg tablets and one 0.75 mg tablet in the morning and one placebo tablet in the evening for 24 weeks. Placebo tablets given to maintain blind.
  Interventions: Drug: Baricitinib; Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104; INCB28050
  Arms: Baricitinib 0.75 mg/0.5 mg BID; Baricitinib 0.75 mg/0.5 mg QD; Baricitinib 1.5 mg/1 mg; Baricitinib 4 mg/2.75 mg
Drug: Placebo — Administered orally

SUMMARY:
This is a dose ranging study to evaluate the safety and efficacy of baricitinib in the treatment of participants with mild to moderate diabetic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Type 2 diabetes treated with at least one antihyperglycemic medicine for 12 months
* Have diabetic kidney disease and receiving one of two specific medicines used to treat high blood pressure or diabetic kidney disease for at least 3 months
* Estimated Glomerular Filtration Rate (eGFR) of 25 to 70 milliliter per minute per 1.73 square meter (mL/min/1.73 m²) (as determined by the Chronic Kidney Disease Epidemiology Collaboration equation) and a urinary albumin/creatinine ratio (UACR) >300 milligram per gram (mg/g) and <5000 mg/g

Exclusion Criteria:

* Too high blood pressure when you enter the study
* Some specific medicines used to treat high blood pressure or diabetic kidney disease
* Frequent high blood glucose levels
* Renal transplant or past history of dialysis
* Nonsteroidal anti-inflammatory drugs (NSAIDs)
* Had a special X-ray in the past 30 days which involved also receiving an injection of dye into the vein
* Major surgery within 8 weeks of study entry or will require major surgery during the study
* Some types of vaccination
* Shingles or currently have symptoms of a cold sore
* Serious viral, bacterial, fungal, or parasitic infection, or a urinary infection, Tuberculosis (TB)
* Human immunodeficiency virus (HIV) infection- the virus that causes Acquired immunodeficiency syndrome (AIDS)
* Have or had some blood disorders, enlarged lymph glands or spleen, or some cancers.
* Serious circulatory, breathing, liver, stomach or bowel problems, neurological or psychiatric disorders
* Heart attack or heart failure, or a stroke
* Other serious disorders or illnesses
* Electrocardiogram (ECG) heart trace abnormalities
* Alcohol or illegal drug abuse
* Donated more than 500 mL of blood in the last 30 days (no blood donations allowed during the study)
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-08; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (44):
- United States (35):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lancaster, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torrance, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lakewood, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Augusta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Meridian, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gurnee, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peoria, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rockville, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ann Arbor, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pontiac, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Billings, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashua, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albany, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosedale, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winston-Salem, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bethlehem, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sumter, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chattanooga, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wenatchee, Washington
- Japan (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ibaraki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mérida
- Puerto Rico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio Piedras

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included a 24-week treatment period and a 4- to 8-week washout period where study drug was discontinued. Time to loss-of-treatment benefit (defined as a failure to maintain a 30% decrease in UACR from baseline) was evaluated at Week 28. Participants who maintained treatment benefit were followed for an additional 4 weeks.
Pre-assignment Details: Participants in each baricitinib dose group were classified by their baseline estimated glomerular filtration rate (eGFR) into higher (50 to 70 milliliter [mL]/minute [min]/1.73 meters squared [m²]) and lower (25 to <50 mL/min/1.73 m²) eGFR strata. Participants in the lower strata had their dose adjusted to a lower dose.
Groups:
- Placebo: Placebo administered orally (PO) once a day (QD).
- Baricitinib 0.75 mg/0.5 mg QD: Baricitinib 0.75 mg or 0.5 mg administered PO QD.
- Baricitinib 0.75 mg/0.5 mg BID: Baricitinib 0.75 mg or 0.5 mg administered PO twice a day (BID).
- Baricitinib 1.5 mg/1 mg: Baricitinib 1.5 mg or 1 mg administered PO QD.
- Baricitinib 4 mg/2.75 mg: Baricitinib 4 milligram (mg) or 2.75 mg administered PO QD.
Period: Treatment Period (Weeks 1-24)
Arm/Group | Placebo | Baricitinib 0.75 mg/0.5 mg QD | Baricitinib 0.75 mg/0.5 mg BID | Baricitinib 1.5 mg/1 mg | Baricitinib 4 mg/2.75 mg
Started | 27 | 25 | 27 | 26 | 25
Received at Least One Dose of Study Drug | 27 | 25 | 26 | 26 | 25
Completed | 27 | 21 | 26 | 24 | 23
Not Completed | 0 | 4 | 1 | 2 | 2
Not completed — Inappropriately Enrolled | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 3 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1
Period: Washout Period 1 (Weeks 25-28)
Arm/Group | Placebo | Baricitinib 0.75 mg/0.5 mg QD | Baricitinib 0.75 mg/0.5 mg BID | Baricitinib 1.5 mg/1 mg | Baricitinib 4 mg/2.75 mg
Started | 27 | 21 | 26 | 24 | 23
Completed | 24 | 17 | 25 | 22 | 20
Not Completed | 3 | 4 | 1 | 2 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 4 | 0 | 1 | 2
Period: Washout Period 2 (Weeks 29-32)
Arm/Group | Placebo | Baricitinib 0.75 mg/0.5 mg QD | Baricitinib 0.75 mg/0.5 mg BID | Baricitinib 1.5 mg/1 mg | Baricitinib 4 mg/2.75 mg
Started | 6 (Study was completed at Week 28 for 18 participants.) | 6 (Study was completed at Week 28 for 11 participants.) | 8 (Study was completed at Week 28 for 17 participants.) | 6 (Study was completed at Week 28 for 16 participants.) | 12 (Study was completed at Week 28 for 8 participants.)
Completed | 6 | 6 | 7 | 6 | 9
Not Completed | 0 | 0 | 1 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 3
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants that received at least one dose of study drug.
Groups:
- Placebo: Placebo administered PO QD.
- Baricitinib 0.75/0.5 mg QD: Baricitinib 0.75 mg or 0.5 mg administered PO QD.
- Baricitinib 0.75 mg/0.5 mg BID: Baricitinib 0.75 mg or 0.5 mg administered PO BID.
- Baricitinib 1.5 mg/1 mg QD: Baricitinib 1.5 mg or 1 mg administered PO QD.
- Baricitinib 4 mg/2.75 mg: Baricitinib 4 mg or 2.75 administered PO QD.
- Total: Total of all reporting groups
Arm/Group | Placebo | Baricitinib 0.75/0.5 mg QD | Baricitinib 0.75 mg/0.5 mg BID | Baricitinib 1.5 mg/1 mg QD | Baricitinib 4 mg/2.75 mg | Total
Number analyzed (Participants) | 27 | 25 | 26 | 26 | 25 | 129
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64 (9.0) | 61 (10.0) | 64 (8.3) | 61 (10.4) | 63 (7.8) | 63 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 5 | 5 | 10 | 35
  Male | 20 | 17 | 21 | 21 | 15 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 6 | 7 | 4 | 25
  Not Hispanic or Latino | 23 | 21 | 20 | 19 | 21 | 104
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 2 | 2 | 1 | 9
  Asian | 14 | 12 | 12 | 11 | 11 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 2 | 7 | 3 | 0 | 3 | 15
  White | 8 | 4 | 9 | 13 | 9 | 43
  More than one race | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 0 | 1 | 0 | 0 | 0 | 1
  United States | 14 | 13 | 14 | 14 | 13 | 68
  Japan | 11 | 10 | 10 | 10 | 11 | 52
  Mexico | 2 | 1 | 2 | 2 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Urinary Albumin/Creatinine Ratio (UACR) at Week 24
Description: UACR is a potential marker of chronic kidney disease, calculated as a ratio of Urinary Albumin and Urinary Creatinine. The least squares mean (LS mean) are from mixed model repeated measures (MMRM) analyses which include treatment, baseline estimated Glomerular Filtration Rate (eGFR) group (higher: 50 to 70 mL/min/1.73m² and lower: 25 to <50 mL/min/1.73m²), visit, treatment-by-visit interaction, baseline UACR, and baseline UACR-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: milligram/gram (mg/g)
Groups:
- Baricitinib 4 mg/2.75 mg: Baricitinib 4 mg or 2.75 mg administered PO QD.
Arm/Group | Placebo | Baricitinib 0.75 mg/0.5 mg QD | Baricitinib 0.75 mg/0.5 mg BID | Baricitinib 1.5 mg/1 mg | Baricitinib 4 mg/2.75 mg
Number analyzed (Participants) | 27 | 25 | 26 | 26 | 25
milligram/gram (mg/g) | 1.12 (0.172) | 0.87 (0.155) | 0.85 (0.131) | 0.91 (0.143) | 0.66 (0.111)

2. Secondary Outcome: Change From Baseline in Urinary Monocyte Chemotactic Protein 1 (MCP-1)/Creatinine Ratio
Time Frame: Baseline, Week 24
Population: Zero participants analyzed. No data analyzed due to urinary MCP-1 and creatinine being measured on different urine samples from different time points and thus not able to correlate.
Arm/Group | Placebo | Baricitinib 0.75 mg/0.5 mg QD | Baricitinib 0.75 mg/0.5 mg BID | Baricitinib 1.5 mg/1 mg | Baricitinib 4 mg/2.75 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in Creatinine Clearance at Week 24
Description: Creatinine clearance is the amount of creatinine cleared from kidney within 24 hours. The LS mean was from MMRM analyses which included treatment, baseline eGRF group, visit, treatment-by-visit interaction, baseline Creatinine Clearance, and baseline Creatinine Clearance-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: milliliter/minute (mL/min)
Arm/Group | Placebo | Baricitinib 0.75 mg/0.5 mg QD | Baricitinib 0.75 mg/0.5 mg BID | Baricitinib 1.5 mg/1 mg | Baricitinib 4 mg/2.75 mg
Number analyzed (Participants) | 27 | 25 | 26 | 26 | 25
milliliter/minute (mL/min) | 0.93 (0.070) | 1.09 (0.104) | 0.86 (0.069) | 0.86 (0.069) | 0.080 (0.066)

4. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) at Week 24
Description: EQ-5D-5L is a 2-part measurement. The first part is comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive the health state index scores using the United Kingdom (UK) algorithm, with scores ranging from -0.594 to 1, and the United States (US) algorithm, with scores ranging from -0.109 to 1. A higher score indicates better health state. The second part is assessed using a visual analog scale (VAS) that ranged from 0 to 100mm, where 0 is the worst health you can imagine and 100 is the best health you can imagine. The LS means are analyzed using an analysis of covariance (ANCOVA) model with treatment, baseline eGFR group, and baseline VAS score or baseline health state index score as covariates.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least one dose of study drug. Missing values were imputed with the last observation carried forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Baricitinib 0.75 mg/0.5 mg QD | Baricitinib 0.75 mg/0.5 mg BID | Baricitinib 1.5 mg/1 mg | Baricitinib 4 mg/2.75 mg
Number analyzed (Participants) | 27 | 25 | 26 | 26 | 25
Units on a Scale
  Index Score (UK Algorithm) Week 24 | 0.00 (0.03) | -0.03 (0.03) | -0.01 (0.03) | -0.04 (0.03) | 0.00 (0.03)
  Index Score (US Algorithm) Week 24 | 0.00 (0.02) | -0.03 (0.02) | 0.00 (0.02) | -0.03 (0.02) | 0.00 (0.02)
  Self-Perceived Health Score | 2.62 (2.94) | -1.97 (3.02) | 0.28 (2.95) | -5.66 (2.96) | 0.37 (3.02)

5. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration-Time Curve at Steady State (AUC,ss)
Description: Evaluable pharmacokinetic concentrations from the 2-week, 4-week, 8-week, 12-week, 16-week, 20-week and 24-week time points were combined and utilized in a population approach to determine the population mean estimate and standard deviation at steady-state.
Time Frame: Weeks 2 and 4 (1-2 hours postdose), 8 (3-6 hours postdose), 12 (in fasted state), 16 and 20 (6-9 hours postdose), 24 (in fasted state)
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: nanomole*hour (nM*hr)
Arm/Group | Baricitinib 0.75 mg/0.5 mg QD | Baricitinib 0.75 mg/0.5 mg BID | Baricitinib 1.5 mg/1 mg | Baricitinib 4 mg/2.75 mg
Number analyzed (Participants) | 24 | 26 | 26 | 25
nanomole*hour (nM*hr) | 198 (89.9) | 286 (92.4) | 388 (151) | 1250 (577)

ADVERSE EVENTS:
Groups:
- Placebo - Washout 1; Placebo Washout 2: Placebo administered PO QD.
- Baricitinib 0.75 mg/0.5 mg QD - Washout 1; Baricitinib 0.75 mg/0.5 mg QD - Washout 2: Baricitinib 0.75 mg or 0.5 mg administered PO QD.
- Baricitinib 0.75 mg/0.5 mg BID - Washout 1; Baricitinib 0.75 mg/0.5 mg BID - Washout 2: Baricitinib 0.75 mg or 0.5 mg administered PO BID.
- Baricitinib 1.5 mg/1 mg - Washout 1; Baricitinib 1.5 mg/1 mg - Washout 2: Baricitinib 1.5 mg or 1 mg administered PO QD.
- Baricitinib 4 mg/2.75 mg - Washout 1; Baricitinib 4 mg/2.75 mg - Washout 2: Baricitinib 4 mg or 2.75 mg administered PO QD.
Arm/Group | Placebo | Baricitinib 0.75 mg/0.5 mg QD | Baricitinib 0.75 mg/0.5 mg BID | Baricitinib 1.5 mg/1 mg | Baricitinib 4 mg/2.75 mg | Placebo - Washout 1 | Baricitinib 0.75 mg/0.5 mg QD - Washout 1 | Baricitinib 0.75 mg/0.5 mg BID - Washout 1 | Baricitinib 1.5 mg/1 mg - Washout 1 | Baricitinib 4 mg/2.75 mg - Washout 1 | Placebo Washout 2 | Baricitinib 0.75 mg/0.5 mg QD - Washout 2 | Baricitinib 0.75 mg/0.5 mg BID - Washout 2 | Baricitinib 1.5 mg/1 mg - Washout 2 | Baricitinib 4 mg/2.75 mg - Washout 2
Serious Adverse Events (participants affected / at risk) | 2/27 | 0/25 | 2/26 | 2/26 | 6/25 | 0/27 | 0/21 | 0/26 | 0/24 | 0/23 | 0/6 | 0/6 | 1/8 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 18/27 | 18/25 | 17/26 | 19/26 | 23/25 | 5/27 | 4/21 | 4/26 | 7/24 | 8/23 | 1/6 | 2/6 | 1/8 | 0/6 | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=27) | Baricitinib 0.75 mg/0.5 mg QD (N=25) | Baricitinib 0.75 mg/0.5 mg BID (N=26) | Baricitinib 1.5 mg/1 mg (N=26) | Baricitinib 4 mg/2.75 mg (N=25) | Placebo - Washout 1 (N=27) | Baricitinib 0.75 mg/0.5 mg QD - Washout 1 (N=21) | Baricitinib 0.75 mg/0.5 mg BID - Washout 1 (N=26) | Baricitinib 1.5 mg/1 mg - Washout 1 (N=24) | Baricitinib 4 mg/2.75 mg - Washout 1 (N=23) | Placebo Washout 2 (N=6) | Baricitinib 0.75 mg/0.5 mg QD - Washout 2 (N=6) | Baricitinib 0.75 mg/0.5 mg BID - Washout 2 (N=8) | Baricitinib 1.5 mg/1 mg - Washout 2 (N=6) | Baricitinib 4 mg/2.75 mg - Washout 2 (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=27) | Baricitinib 0.75 mg/0.5 mg QD (N=25) | Baricitinib 0.75 mg/0.5 mg BID (N=26) | Baricitinib 1.5 mg/1 mg (N=26) | Baricitinib 4 mg/2.75 mg (N=25) | Placebo - Washout 1 (N=27) | Baricitinib 0.75 mg/0.5 mg QD - Washout 1 (N=21) | Baricitinib 0.75 mg/0.5 mg BID - Washout 1 (N=26) | Baricitinib 1.5 mg/1 mg - Washout 1 (N=24) | Baricitinib 4 mg/2.75 mg - Washout 1 (N=23) | Placebo Washout 2 (N=6) | Baricitinib 0.75 mg/0.5 mg QD - Washout 2 (N=6) | Baricitinib 0.75 mg/0.5 mg BID - Washout 2 (N=8) | Baricitinib 1.5 mg/1 mg - Washout 2 (N=6) | Baricitinib 4 mg/2.75 mg - Washout 2 (N=12)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 7 (7) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0
Cardiac hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal sensation in eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0
Injection site nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection parasitic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 (1) | 4 (6) | 4 (4) | 4 (4) | 3 (4) | 0 | 0 | 0 | 0 | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urethritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Occult blood (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Occult blood positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Red blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0
Osteochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head banging (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic bullosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Microscopic polyangiitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days